CLINICAL TRIAL: NCT00003102
Title: Phase I/II Study of 131I-Labeled Chimeric Antibody G250 (131I-cG250) in Patients With Advanced Renal Carcinoma
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065834; MSKCC-97049 (Other: Memorial Sloan-Kettering Cancer Center); NCI-H97-0004 (Other: NCI); LUD 96-006 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 50cGy radiation (Experimental): On day 1, patients received a single dose of 131I-cG250 (5 mCi/5 mg) administered as an intravenous infusion over 10 minutes.
  Therapeutic doses of 131I-cG250 were administered the following week as fractionated outpatient doses, starting with 30 millicurie (mCi)/5 mg 131I-cG250. Subsequent doses of 131I-cG250 were administered at 2-3 day intervals with the total amount of 131I-cG250 administered based on the calculated clearance of the initial dose administered on day 1. Whole body activity was maintained at no more than 30 mCi iodine-131.
  In the absence of disease progression and after recovery from toxicity, patients could be re-treated beginning 8 weeks after the last treatment of the initial series, for a total of not more than 3 treatments.
  Interventions: Biological: Iodine-131 radiolabeled chimeric monoclonal antibody G250 (131I-cG250)
- Cohort 2 75cGy radiation (Experimental): On day 1, patients received a single dose of 131I-cG250 (5 mCi/5 mg) administered as an intravenous infusion over 10 minutes.
  Therapeutic doses of 131I-cG250 were administered the following week as fractionated outpatient doses, starting with 30 millicurie (mCi)/5 mg 131I-cG250. Subsequent doses of 131I-cG250 were administered at 2-3 day intervals with the total amount of 131I-cG250 administered based on the calculated clearance of the initial dose administered on day 1. Whole body activity was maintained at no more than 30 mCi iodine-131.
  In the absence of disease progression and after recovery from toxicity, patients could be re-treated beginning 8 weeks after the last treatment of the initial series, for a total of not more than 3 treatments.
  Interventions: Biological: Iodine-131 radiolabeled chimeric monoclonal antibody G250 (131I-cG250)
- Cohort 3 100cGy radiation (Experimental): On day 1, patients received a single dose of 131I-cG250 (5 mCi/5 mg) administered as an intravenous infusion over 10 minutes.
  Therapeutic doses of 131I-cG250 were administered the following week as fractionated outpatient doses, starting with 30 millicurie (mCi)/5 mg 131I-cG250. Subsequent doses of 131I-cG250 were administered at 2-3 day intervals with the total amount of 131I-cG250 administered based on the calculated clearance of the initial dose administered on day 1. Whole body activity was maintained at no more than 30 mCi iodine-131.
  In the absence of disease progression and after recovery from toxicity, patients could be re-treated beginning 8 weeks after the last treatment of the initial series, for a total of not more than 3 treatments.
  Interventions: Biological: Iodine-131 radiolabeled chimeric monoclonal antibody G250 (131I-cG250)

INTERVENTIONS:
Biological: Iodine-131 radiolabeled chimeric monoclonal antibody G250 (131I-cG250) — cG250 is an IgG1 chimeric monoclonal antibody. It was supplied as a sterile solution at a concentration of 1.0 mg/mL in either a 2 mL or a 5 mL vial. cG250 was radiolabeled with Iodine-131 prior to use.

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of monoclonal antibody therapy in treating patients with advanced kidney cancer.

DETAILED DESCRIPTION:
This is a dose-escalation study. Initially patients receive a scout dose of iodine-131 radiolabeled chimeric monoclonal antibody G250 (131I-cG250) administered intravenously (IV) over 10 minutes to determine whole body clearance. One week later, patients receive incremental doses of 131I-cG250 IV over 10 minutes at 2-3 day intervals for 2-6 weeks,. Dose escalation begins at least 8 weeks after the last infusion of 131I-cG250. In the absence of dose-limiting toxicity in the first 3 patients treated, subsequent cohorts of 3 patients each receive escalating doses of 131I-cG250 on the same schedule. If dose-limiting toxicity occurs in 2 of 6 patients treated at a given dose level, then dose escalation ceases and the next lower dose is declared the maximum tolerated dose (MTD). Treatment continues once recovery from all toxic effects occurs, beginning 8 to 12 weeks following the last dose of 131I-cG250. Patients achieving complete remission, partial remission, or stable disease were eligible to receive up to 3 courses of treatment.

ELIGIBILITY:
Inclusion Criteria

Histologically proven renal cell carcinoma. Clinical presentation consistent with metastatic renal cell carcinoma. Bidimensionally measurable disease by conventional imaging. Patients must have been off chemotherapy or immunotherapy for at least 6 weeks prior to study entry.

Women of child-bearing age must have had a negative pregnancy test carried out the day of and prior to receiving therapy, and were asked to use effective contraception during the study.

Patients were required to be ambulatory with a Karnofsky Performance Status at least 70, Serum creatinine ≤ 2mg/dl, Serum bilirubin ≤ 1mg/d, White Blood Cells (WBC) ≥ 3,500/mm^3, Platelet count ≥ 100,000/mm^3, Prothrombin time < 1.3 x control.

Exclusion Criteria

Significant prior radiation therapy to the entire pelvis and/or lumbosacral spine.

Clinically significant cardiac disease. Serious infection requiring treatment with antibiotics, or other serious illness.

Women who are pregnant or lactating. Central Nervous System (CNS) tumor involvement. Life expectancy less than 6 weeks. Hypercalcemia greater than 12.5 mg/dL or symptomatic.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1998-11-17 (Actual); Primary Completion 2000-04-19 (Actual); Study Completion 2003-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitanya R. Divgi, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 50cGy Radiation; Cohort 2 75cGy Radiation; Cohort 3 100cGy Radiation: On day 1, patients received a single dose of 131I-cG250 (5 mCi/5 mg) administered as an intravenous infusion over 10 minutes.
  Therapeutic doses of 131I-cG250 were administered the following week as fractionated outpatient doses, starting with 30 mCi/5 mg 131I-cG250. Subsequent doses of 131I-cG250 were administered at 2-3 day intervals with the total amount of 131I-cG250 administered based on the calculated clearance of the initial dose administered on day 1. Whole body activity was maintained at no more than 30 mCi iodine-131.
  In the absence of disease progression and after recovery from toxicity, patients could be re-treated beginning 8 weeks after the last treatment of the initial series, for a total of not more than 3 treatments.
  Iodine-131 radiolabeled chimeric monoclonal antibody G250 (131I-cG250): cG250 is an IgG1 chimeric monoclonal antibody. It was supplied as a sterile solution at a concentration of 1.0 mg/mL in either a 2 mL or a 5 mL vial. cG250 was radiolabeled with Iodine-131 prior to use.
Period: Overall Study
Arm/Group | Cohort 1 50cGy Radiation | Cohort 2 75cGy Radiation | Cohort 3 100cGy Radiation
Started | 3 | 9 | 3
Completed | 2 | 6 | 1
Not Completed | 1 | 3 | 2
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Progressive Disease | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 50cGy Radiation: On day 1, patients received a single dose of 131I-cG250 (5 mCi/5 mg) administered as an intravenous infusion over 10 minutes.
  Therapeutic doses of 131I-cG250 were administered the following week as fractionated outpatient doses, starting with 30 mCi/5 mg 131I-cG250. Subsequent doses of 131I-cG250 were administered at 2-3 day intervals with the total amount of 131I-cG250 administered based on the calculated clearance of the initial dose administered on day 1. Whole body activity was maintained at no more than 30 mCi iodine-131.
  In the absence of disease progression and after recovery from toxicity, patients could be re-treated beginning 8 weeks after the last treatment of the initial series, for a total of not more than 3 treatments.
  Iiodine-131 radiolabeled chimeric monoclonal antibody G250 (131I-cG250): cG250 is an IgG1 chimeric monoclonal antibody. It was supplied as a sterile solution at a concentration of 1.0 mg/mL in either a 2 mL or a 5 mL vial. cG250 was radiolabeled with Iodine-131 prior to use.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 50cGy Radiation | Cohort 2 75cGy Radiation | Cohort 3 100cGy Radiation | Total
Number analyzed (Participants) | 3 | 9 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 2 | 13
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 2 | 8 | 1 | 11
Region of Enrollment [Number; unit: participants]
  United States | 3 | 9 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs)
Description: All adverse events occurring during the study were to be recorded on the patient's case report form, and include the following information: a description; date of onset and resolution; severity; relationship to an investigational agent; action taken and outcome. Toxicity was graded in accordance with the NCI CTCAE version 3.0.
Time Frame: Up to 12 months
Population: All patients who received at least one dose of 131I-cG250.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 50cGy Radiation | Cohort 2 75cGy Radiation | Cohort 3 100cGy Radiation
Number analyzed (Participants) | 3 | 9 | 3
Participants | 3 | 8 | 3

2. Primary Outcome: Number of Patients With Dose-Limiting Toxicities (DLTs)
Description: Subjects were monitored for Adverse Events (AEs) for at least 8 weeks after the last infusion of 131I-cG250, or until recovery from all toxicity, and prior to dose escalation. Toxicity was graded in accordance with the Common Toxicity Criteria (CTC) of the National Cancer Institute (NCI) Version 3.0. Dose-Limiting Toxicity (DLT) was defined as grade 3 or greater toxicity related to study therapy. The maximum tolerated dose was defined as the highest safely tolerated dose where at most one of six patients experiences a DLT with the next higher dose having at least two patients who experience a DLT.
Time Frame: up to 12 months
Population: All patients who received at least one dose of 131I-cG250.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 50cGy Radiation | Cohort 2 75cGy Radiation | Cohort 3 100cGy Radiation
Number analyzed (Participants) | 3 | 9 | 3
Participants | 0 | 1 | 3

3. Secondary Outcome: Number of Patients With Best Overall Tumor Response
Description: Tumor responses were evaluated using computed tomography and categorized according to World Health Organization (WHO) criteria at baseline and at no more than 6 weeks after the last dose, or not more than 12 weeks after entry into the study. Complete Response (CR): disappearance of all measurable disease lasting at least 1 month; Partial Response (PR): ≥ 50% decrease in the size of the product of 2 perpendicular diameters of any measurable lesions and no new lesions, lasting at least one month; Progressive Disease (PD): ≥ 25% increase in the size of any measurable lesions or the appearance of any new lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 12 weeks
Population: All patients who received study treatment and had at least one pre- and post-treatment tumor measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 50cGy Radiation | Cohort 2 75cGy Radiation | Cohort 3 100cGy Radiation
Number analyzed (Participants) | 3 | 7 | 2
Participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0
  Stable Disease (SD) | 2 | 6 | 1
  Progressive Disease (PD) | 1 | 1 | 1

4. Secondary Outcome: Number of Patients With Human Anti-chimeric Antibodies (HACA)
Description: Blood samples were taken at baseline and in weeks 2, 3, 4, 5, and 6 as well as month 6. HACA was measured by an enzyme-linked immunosorbent assay (ELISA) using the "double antibody sandwich" technique and pretreatment serum as negative control.
Time Frame: Up to 6 months
Population: All patients who received study therapy and had blood samples taken for HACA analyses before and after treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 50cGy Radiation | Cohort 2 75cGy Radiation | Cohort 3 100cGy Radiation
Number analyzed (Participants) | 3 | 9 | 3
Participants
  Number of subjects with negative HACA before and after treatment | 2 | 8 | 3
  Number of subjects with negative HACA before treatment and positive HACA after treatment | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: up to 12 months
Description: All adverse events occurring during the study were to be recorded on the patient's case report form, and include the following information: a description; date of onset and resolution; severity; relationship to an investigational agent; action taken and outcome. Toxicity was graded in accordance with the NCI CTCAE version 3.0.
Arm/Group | Cohort 1 50cGy Radiation | Cohort 2 75cGy Radiation | Cohort 3 100cGy Radiation
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/9 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/9 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 8/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 50cGy Radiation (N=3) | Cohort 2 75cGy Radiation (N=9) | Cohort 3 100cGy Radiation (N=3)
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 50cGy Radiation (N=3) | Cohort 2 75cGy Radiation (N=9) | Cohort 3 100cGy Radiation (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2
Abdominal distention (Gastrointestinal disorders) | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Faeces discolored (Gastrointestinal disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dysuria (Nervous system disorders) | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Feeling cold (General disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dypsnea (Cardiac disorders) | 2 | 3 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Oedema peripheral (Cardiac disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Heamoptysis (Vascular disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 2
Pyrexia (General disorders) | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Insomnia (Nervous system disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Melena (Gastrointestinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Herpes zoster (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Taste disorder (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 0
Urinary hemmorhage (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No